CLINICAL TRIAL: NCT03610620
Title: Does Ex-vivo Fluorescence Confocal Microscopy Allow Faster Evaluation of Margin Clearance in Basal Cell Carcinomas in Mohs Surgery: A Pilot Study
Brief Title: Confocal Microscopy Evaluation of Margin Clearance in Basal Cell Carcinomas in Mohs Surgery
Acronym: FCM-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Dawson (Other)
Collaborators: Mavig GmbH (Industry)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 212591
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal cell carcinoma; Mohs surgery; Vivascope 2500 ex-vivo fluorescent confocal microscope; Frozen section Mohs histology
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: Compare accuracy and speed of the Vivascope 2500 to frozen sections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARM A (Experimental): Vivascope 2500 ex-vivo fluorescent confocal microscope
  Interventions: Procedure: Vivascope 2500 ex-vivo fluorescent confocal microscope

INTERVENTIONS:
Procedure: Vivascope 2500 ex-vivo fluorescent confocal microscope — scanned with the Vivascope 2500

SUMMARY:
This study is comparing the accuracy and speed of the Vivascope 2500 ex-vivo fluorescent confocal microscope with frozen section Mohs histology in evaluating clear margins in basal cell carcinoma in Mohs surgery.

DETAILED DESCRIPTION:
Patients with basal cell carcinomas in the head and neck area, being considered for Mohs surgery with frozen sections will be invited to participate in this trial by the investigators when they attend for their pre-surgical consultation. They will be given sufficient time to review the information sheet and ask questions. When they attend for their Mohs surgery, they will be recruited if they wish to participate in this trial, at which point, the investigator, or an authorized member of their team, will obtain written informed consent for patients. The patient will then undergo Mohs surgery. The processing and interpretation with frozen sections will be conducted in the same way, the only difference being immediately after the BCC is excised with a Mohs bevelled edge (45o incision), the tissue is immersed in acridine orange (nuclear DNA stain) and placed upside down with the deep margin of the tissue face up. With a glass slide placed on top, we would place the FCM (Vivascope 2500) over this, scan the tissue and obtain mosaic images of the tissue which would be stitched together. The penetration of the FCM scan is approximately 0.25mm. This is approximately the distance between 2-3 Mohs wafers. The investigators would usually consider a margin of 3 Mohs wafers (300 microns) clear. When the scanning is completed (5 minutes), the Mohs layer would be sent for frozen section (stained with haematoxylin and eosin) for confirmation in the usual way. The Mohs surgeon can interpret the FCM mosaic images later. Acridine orange does not interfere with frozen sections or paraffin histopathological quality. No medicines will be used in this study. The information is collected on only 1 patient visit. There is no follow up period. The main objectives would (1) compare the accuracy in detection of BCC margins with FCM compared with FSM and (2) evaluate the time taken for processing and interpretation of FCM (acridine orange inking and rinsing, image acquisition and mosaic stitching, and image interpretation) compared with the time taken for processing and interpretation of FSM (sample flattening, freezing and cutting with the cryostat, H&E staining, slide cover slipping and slide interpretation).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patient with basal cell carcinoma on the head and neck undergoing Mohs surgery with frozen sections
3. Patient willing and able to give informed consent
4. Patient treated not previously or currently treated with a hedgehog inhibitor medication (vismodegib)
5. Patient suitable for Mohs surgery
6. Excised lesion suitable for scanning with FCM as determined by investigator -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
To compare the specificity and sensitivity of the ex-vivo fluorescence confocal microscopy against frozen section histopathology in detecting residual BCC in Mohs excisions. | 1 DAY
  Compare the specificity and sensitivity of the ex-vivo fluorescence confocal microscopy against frozen section histopathology in detecting residual BCC in Mohs excisions.

SECONDARY OUTCOMES:
To compare the time taken for processing and interpretation of the ex-vivo fluorescence confocal microscopy against frozen section histopathology in detecting residual BCC in Mohs excisions. | 1 DAY
  Compare the time taken for processing and interpretation of the ex-vivo fluorescence confocal microscopy against frozen section histopathology in detecting residual BCC in Mohs excisions.

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Tan, Consultant, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK)
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom